CLINICAL TRIAL: NCT02289157
Title: Negative Pressure Wound Therapy in High Risk Patients Undergoing Cesarean
Brief Title: Negative Pressure Wound Therapy in Cesarean Section
Acronym: NPWTCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: KCI USA, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU 042014-047
Record Dates: First submitted 2014-10-06; First posted 2014-11-13 (Estimated); Results first posted 2018-07-02 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2018-05

CONDITIONS: Postoperative Wound Complications
MeSH Terms: interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Intervention Model Description: Randomized Placebo Controlled Clinical Trial - Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Negative Pressure Wound Therapy (Experimental): After standard cesarean section completed patients will have Prevena negative pressure wound therapy system placed.
  Interventions: Device: Negative pressure wound therapy
- Standard dressing (No Intervention): After standard cesarean section completed patients will have standard dressing placed.

INTERVENTIONS:
Device: Negative pressure wound therapy — Single use negative pressure wound therapy systems are composed of a pressure pump and dressing kit. The pump creates a negative pressure of 125 mmHg (+/- 20 mgHg) and the dressing directly covers surgical incision. The system is battery-powered and designed to be used for a minimum of two days and a maximum of seven days of continuous use. The investigators hypothesize that negative pressure wound therapy will decrease the wound complications in these patients. The investigators will be using Prevena Incision Management System as the negative pressure device in our study.
  Other Names: Prevena
  Arms: Negative Pressure Wound Therapy

SUMMARY:
The investigators propose a prospective, randomized trial evaluating the use of negative pressure wound therapy (NPWT) with high risk obstetrical patients. The investigators hypothesize that negative pressure wound therapy will decrease the wound complications in these patients. The investigators aim to look at all wound complications such as infection and disruption and will be using Prevena incision management system for our NPWT device .

DETAILED DESCRIPTION:
This will be a prospective, randomized, controlled trial of pregnant women who present for prenatal care at Parkland Health and Hospital System. The participants will be limited to women undergoing a cesarean section who are high risk for wound complications: all patients with a BMI > 40 undergoing cesarean section.

The primary outcome will be wound complication defined as wound disruption or wound infection. A wound disruption will be defined as the partial or complete opening of the deep subcutaneous space, not to include superficial skin separation. Underlying causes will include seroma, hematoma, abscess, and facial dehiscence. Wound infection will be defined as a physician diagnosis of wound infection with erythema and warmth extending beyond the immediate area adjacent to the incision and requiring treatment with antibiotics.

All patients with a BMI > 40 undergoing scheduled cesarean section and patients with a BMI >40 who are admitted in labor will be approached to participate in the study. If patients meeting this criteria undergo cesarean section, they will be randomized to negative pressure wound therapy or a standard dressing. All labor treatment, pre-operative antibiotics, surgical technique, and post-operative care will not differ from current standard of care. All patients randomized will be included in the study.

All study participants will have the thickness of their subcutaneous tissue measured with a sterile ruler. Patients randomized to NPWT will have a negative pressure wound therapy system placed over her incision per the manufacturer's protocol. All patients randomized to standard dressing will have the customary dressing of gauze and surgical tape placed over her incision.

The investigators will be utilizing a single use negative pressure wound therapy system for the study. Single use negative pressure wound therapy systems are composed of a pressure pump and dressing kit. The pump creates a negative pressure of 125 mmHg (+/- 20 mgHg) and the dressing directly covers surgical incision. The system is battery-powered and designed to be used for a minimum of two days and a maximum of seven days of continuous use.

All randomized patients will undergo an examination of their incision by a research physician or nurse prior to discharge. The NPWT will be removed prior to discharge or on post-operative day seven, whichever comes first. All postpartum patients who undergo a cesarean delivery are inpatients until at least post-operative day three and will continue use of NPWT until day of discharge. In patients randomized to a standard dressing, the dressing will be removed prior to discharge per current standard of care.

All randomized patients will also undergo a 2 week post-operative incisional examination by a research physician or nurse at the obstetrical complications clinic. Patients will be followed until 30 days postpartum for any wound complications to include wound infection (superficial and deep), readmission to the hospital, re-operation for wound complications, hematoma, seroma, dehiscence, superficial infection requiring antibiotics, or additional clinical evaluations for wound care in the emergency room or clinic setting. A research physician or nurse will contact each after at least 30 days post-operative to confirm the patients' status and ensure no evaluations, admissions, or interventions were done at outside facilities.

Subjects will exit the study if they are unable to complete the post-operative visit or withdrawal consent for participation.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with BMI > 40 undergoing a cesarean delivery at Parkland Health and Hospital System.

Exclusion Criteria:

* Any patient not meeting inclusion criteria will be deemed ineligible.
* All HIV positive patients will be excluded due to the increased risk of infectious complications in these patients.
* Although patients on anticoagulants can use NPWT, they will be excluded as there may be an increased risk of bleeding in these patients.
* according to the wound therapy manufacturer's instructions patients with:

  * fragile skin
  * allergy to silver or acrylic adhesives
  * a malignancy in the wound bed or margins of the wound bed
  * non-enteric and unexplored fistulas
  * necrotic tissue with eschar present
  * exposed arteries, veins, nerves or organs, anastomotic sites, or surgical suction are not candidates for usage of the device.

Ages: 10 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 441 (Actual)
Dates: Start 2015-01-27 (Actual); Primary Completion 2016-08-30 (Actual); Study Completion 2016-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Roberts, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Parkland Memorial Hospital, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hussamy DJ, Wortman AC, McIntire DD, Leveno KJ, Casey BM, Roberts SW. Closed Incision Negative Pressure Therapy in Morbidly Obese Women Undergoing Cesarean Delivery: A Randomized Controlled Trial. Obstet Gynecol. 2019 Oct;134(4):781-789. doi: 10.1097/AOG.0000000000003465. PMID 31503147

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited in the Parkland Hospital Maternal-Fetal Medicine High Risk Clinic, on the Antepartum Floor, in Labor and Delivery, and in the preoperative holding area. January 2015 until July 2016. 850 screened. See Figure 1 Flow Diagram.
Pre-assignment Details: Patients were excluded for pre-specified exclusion criteria and if they delivered vaginally after consent was obtained. 850 patients were screened. 173 declined participation, 5 withdrew consent, 2 delivered at outside facility, 211 delivered vaginally, 10 did not meet inclusion criteria, and 8 not identified to be enrolled.
Period: Overall Study
Arm/Group | Negative Pressure Wound Therapy | Standard Dressing
Started | 222 | 219
No Post op Check or Follow up Phone Call | 2 | 4
Completed | 222 | 219
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Negative Pressure Wound Therapy | Standard Dressing | Total
Number analyzed (Participants) | 222 | 219 | 441
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.1 (6.1) | 30.3 (6.1) | 29.7 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 222 | 219 | 441
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Race Black | 56 | 60 | 116
  Race Hispanic | 151 | 146 | 297
  Race White | 15 | 13 | 28
Gestational age at delivery [Mean (Standard Deviation); unit: weeks] | 38.6 (1.9) | 38.7 (4.5) | 38.6 (3.5)
Parity [Number; unit: participants] — Number of deliveries after 20 weeks prior to the present delivery
  participants
    Parity 0 | 55 | 42 | 97
    Parity 1 | 64 | 68 | 132
    Parity 2 | 62 | 57 | 119
    Parity > 2 | 41 | 52 | 93
BMI at Delivery [Mean (Standard Deviation); unit: BMI = kg/meter^2] | 46.6 (6.0) | 45.8 (5.8) | 46.3 (6.2)
Tobacco use [Number; unit: participants] — Number of smokers in each arm numbers
  participants | 18 | 15 | 33
Chronic hypertension [Number; unit: participants] | 40 | 36 | 76
Insulin Requiring Diabetes [Number; unit: participants] | 36 | 24 | 60
Primary Cesarean [Number; unit: participants] | 95 | 80 | 175
Cesarean Priority [Number; unit: participants]
  Scheduled | 72 | 72 | 144
  ASAP | 141 | 138 | 279
  Emergent | 9 | 9 | 18
Length of Surgery [Median (Inter-Quartile Range); unit: minutes] | 84 [70 to 103] | 80 [64 to 99] | 82 [67 to 101]
Estimated blood loss [Mean (Standard Deviation); unit: ml] | 1181 (294) | 1136 (285) | 1159 (291)
Midline skin incision [Number; unit: participants] | 170 | 158 | 328
Suture skin closure [Count of Participants; unit: Participants] | 210 | 211 | 421
Subcutaneous skin depth in cm [Mean (Standard Deviation); unit: cm] | 5.5 (1.3) | 5.3 (1.8) | 5.4 (1.7)
Number subcutaneous layers closed [Median (Inter-Quartile Range); unit: layers] | 3 [2 to 4] | 3 [2 to 4] | 3 [2 to 4]
Incision length in cm [Mean (Standard Deviation); unit: cm] | 14.5 (2.5) | 14.6 (2.9) | 14.6 (2.7)
Patients in labor prior cesarean [Count of Participants; unit: Participants] | 44 | 32 | 76
Induction Labor [Count of Participants; unit: Participants] | 47 | 43 | 90
Ruptured Membranes [Count of Participants; unit: Participants] | 77 | 59 | 136
Chorioamnionitis [Count of Participants; unit: Participants] | 15 | 12 | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Wound Complication
Description: Number of Patients with Wound infection complications: hematoma, seroma, dehiscence, or Surgical Site Infection.
Time Frame: Day of surgery to 30 days postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Negative Pressure Wound Therapy | Standard Dressing
Number analyzed (Participants) | 222 | 219
Participants | 37 | 42
Statistical Analysis 1: Comparison: Negative Pressure Wound Therapy vs Standard Dressing; Test type: Other; p = 0.54, Regression, Logistic; Ho: There is no difference between number of patients with wound complications between the study (icNPT) and comparison groups; Risk Ratio (RR) = 0.9, 95% CI 2-sided [0.5 to 1.4]

2. Primary Outcome: Number of Participants With Classification of Wound Morbidity
Description: Listing of different types of wound morbidity in the 2 cohorts: dehiscence, cellulitis, superficial SSI, deep SSI, organ space SSI
Time Frame: Day of Surgery to 30 days postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Negative Pressure Wound Therapy | Standard Dressing
Number analyzed (Participants) | 222 | 219
Participants
  Dehiscence | 4 | 1
  Cellulitis | 12 | 16
  Superficial incisional SSI | 20 | 25
  Deep incisional SSI | 0 | 0
  Organ space infection | 1 | 0
Statistical Analysis 1: Comparison: Negative Pressure Wound Therapy vs Standard Dressing; Ho: There is no difference between the types wound morbidity in the study (icNPT) and comparison groups; Test type: Other; p = 0.31, Chi-squared; Pearson Chi-squared, df (3)

3. Secondary Outcome: Length of Postoperative Stay
Description: Number of Days in Hospital after Initial Surgery
Time Frame: Length of Postoperative Stay
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Negative Pressure Wound Therapy | Standard Dressing
Number analyzed (Participants) | 222 | 219
days | 3 [3 to 4] | 3 [3 to 4]
Statistical Analysis 1: Comparison: Negative Pressure Wound Therapy vs Standard Dressing; Test type: Other; p = 0.54, Wilcoxon (Mann-Whitney) — Ho: There is no difference between initial length of stay between the study (icNPT) and comparison groups

4. Secondary Outcome: Length of Stay After Readmission
Description: Number of days in hospital after readmission for wound morbidity
Time Frame: After dismissal and readmitted within 30 days for wound morbidity
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Negative Pressure Wound Therapy | Standard Dressing
Number analyzed (Participants) | 222 | 219
days | 16 [6 to 22] | 21 [11 to 25]
Statistical Analysis 1: Comparison: Negative Pressure Wound Therapy vs Standard Dressing; Ho: There is no difference in length of stay after readmission for wound morbidity between the study (icNPT) and comparison groups; Test type: Other; p = 0.41, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Number of Patients With Emergency Room Visits After Discharge
Description: Number of emergency room visits made after initial discharge by the study (icNPT) and comparison groups.
Time Frame: Day of surgery to 30 days postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Negative Pressure Wound Therapy | Standard Dressing
Number analyzed (Participants) | 222 | 219
Participants
  No ER visits | 190 | 190
  1 ER visit | 30 | 28
  2 ER visits | 2 | 1
Statistical Analysis 1: Comparison: Negative Pressure Wound Therapy vs Standard Dressing; Ho: There is no difference between the number of ER visits made per person between the study (icNPT) and comparison groups; Test type: Other; p = 0.38, Chi-squared

6. Secondary Outcome: Number of Patients With Number of Clinic Visits
Description: Number of clinic visits made by patients after surgery concerning wound morbidity per patient
Time Frame: Day of surgery to 30 days postoperative
Measure: Number; unit: participants
Arm/Group | Negative Pressure Wound Therapy | Standard Dressing
Number analyzed (Participants) | 222 | 219
participants
  1 visit | 15 | 15
  2 visits | 4 | 6
  3 visits | 5 | 2
  4 visits | 1 | 4
  5 visits | 1 | 0
Statistical Analysis 1: Comparison: Negative Pressure Wound Therapy vs Standard Dressing; Test type: Other; p = 0.48, Chi-squared — Ho: There is no difference between the number of visits made to the clinic for wound morbidity per patient between the study (icNPT) and comparison groups

7. Secondary Outcome: Number of Participants With Morbid Outcomes After Delivery
Time Frame: Day of Surgery to 30 days postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Negative Pressure Wound Therapy | Standard Dressing
Number analyzed (Participants) | 222 | 219
Participants
  Readmission | 12 | 9
  Postoperative antimicrobials | 33 | 39
  Reoperation for I and D/Extirpation | 14 | 10
Statistical Analysis 1: Comparison: Negative Pressure Wound Therapy vs Standard Dressing; Ho: There is no difference between number of readmissions between the study (icNPT) and comparison groups; Test type: Other; p = 0.52, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Negative Pressure Wound Therapy vs Standard Dressing; Ho: There is no difference in the use of post operative antimicrobials between the the study (icNPT) and comparison groups; Test type: Other; p = 0.45, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Negative Pressure Wound Therapy vs Standard Dressing; Ho: There is no difference in the number of patients with Incision and Drainage and/or Extirpation between the study (icNPT) and comparison groups; Test type: Other; p = 0.44, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Number of Participants With Scheduled and Unscheduled Cesarean Section
Description: Cochran Mantel-Hanzel measures used to compare interactions between scheduled and unscheduled cesarean sections stratified by icNPT and standard dressing, for wound morbidity
Time Frame: Day of Surgery to 30 days postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Negative Pressure Wound Therapy | Standard Dressing
Number analyzed (Participants) | 37 | 42
Participants
  Scheduled | 12 | 12
  Unscheduled | 25 | 30
Statistical Analysis 1: Comparison: Negative Pressure Wound Therapy vs Standard Dressing; Test type: Other — Cochran-Mantel-Haenzel test for interactions between different risk factors: scheduled vs unscheduled cesarean section and icNPT vs Standard dressing; p = 0.68, Cochran-Mantel-Haenszel — Ho: There is no difference between patients with wound morbidity that is significantly affected by the use of icNPT and whether or not the cesarean is scheduled or unscheduled

9. Secondary Outcome: Number of Participants With Pfannenstiel Versus Midline Abdominal Incisions for Cesarian Section
Description: Cochran-Mantel-Haenzel test for interactions between pfannenstiel and midline abdominal incisions stratified by icNPT vs Standard dressing, for wound morbidity
Time Frame: Day of Surgery to 30 days postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Negative Pressure Wound Therapy | Standard Dressing
Number analyzed (Participants) | 37 | 42
Participants
  pfannenstiel | 3 | 8
  midline | 34 | 34
Statistical Analysis 1: Comparison: Negative Pressure Wound Therapy vs Standard Dressing; Test type: Other — Cochran-Mantel-Haenzel test for interactions between different risk factors: pfannenstiel vs midline abdominal incision and icNPT vs Standard dressing; p = 0.27, Cochran-Mantel-Haenszel

10. Secondary Outcome: Number of Patients With Ruptured and Unruptured Membranes Prior to Cesarean Section
Description: Cochran-Mantel-Haenzel measure used to compare interaction in icNPT and Standard dressing stratified by Ruptured vs Unruptured membranes
Time Frame: Day of Surgery to 30 days postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Negative Pressure Wound Therapy | Standard Dressing
Number analyzed (Participants) | 37 | 42
Participants
  Ruptured | 15 | 17
  Unruptured | 22 | 25
Statistical Analysis 1: Comparison: Negative Pressure Wound Therapy vs Standard Dressing; Test type: Other — Cochran-Mantel-Haenzel test for interactions between different risk factors: ruptured vs unruptured membranes and icNPT vs Standard dressing; p = 0.55, Cochran-Mantel-Haenszel

11. Secondary Outcome: Number of Patients in Labor Versus no Labor Prior to Cesarean Section
Description: Cochran-Mantel-Haenzel measure used to compare interaction in icNPT and Standard dressing stratified by patients in labor and patients not in labor
Time Frame: Day of Surgery to 30 days postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Negative Pressure Wound Therapy | Standard Dressing
Number analyzed (Participants) | 37 | 42
Participants
  Labor | 15 | 17
  No labor | 22 | 25
Statistical Analysis 1: Comparison: Negative Pressure Wound Therapy vs Standard Dressing; Test type: Other — Cochran-Mantel-Haenzel test for interactions between labor vs no labor stratified by icNPT vs Standard dressing; p = 0.49, Cochran-Mantel-Haenszel

12. Secondary Outcome: Number of Patients With Hypertension Versus no Hypertension
Description: Cochran-Mantel-Haenzel measure used to compare interaction between patients with hypertension versus no hypertension stratified by icNPT versus standard dressing, in wound morbidity
Time Frame: Day of Surgery to 30 days postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Negative Pressure Wound Therapy | Standard Dressing
Number analyzed (Participants) | 37 | 42
Participants
  Hypertension | 8 | 8
  No Hypertension | 29 | 34
Statistical Analysis 1: Comparison: Negative Pressure Wound Therapy vs Standard Dressing; Test type: Other — Cochran-Mantel-Haenzel measure used to estimate interaction between patients with hypertension versus no hypertension stratified by icNPT versus standard dressing in wound morbidity; p = 0.92, Cochran-Mantel-Haenszel

13. Secondary Outcome: Number of Patients With Insulin Requiring Diabetes Versus no Insulin Requiring Diabetes
Description: Cochran-Mantel-Haenzel measure used to compare interaction in icNPT and Standard wound dressings stratified by women with insulin requiring diabetes and no insulin requiring Diabetes.
Time Frame: Day of Surgery to 30 days postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Negative Pressure Wound Therapy | Standard Dressing
Number analyzed (Participants) | 37 | 42
Participants
  Insulin Diabetes | 5 | 7
  No Diabetes | 32 | 35
Statistical Analysis 1: Comparison: Negative Pressure Wound Therapy vs Standard Dressing; Test type: Other — Cochran-Mantel-Haenzel measure used to estimate interaction in icNPT and Standard wound dressings stratified by women with insulin requiring diabetes and no insulin requiring Diabetes; p = 0.22, Cochran-Mantel-Haenszel

14. Secondary Outcome: Number of Patients With Chorioamnionitis Versus no Chorioamnionitis
Description: Cochran-Mantel-Haenzel measure used to estimate interaction between chorioamnionitis and no chorioamnionitis stratified by icNPT and standard dressing, for wound morbidity
Time Frame: Day of Surgery to 30 days postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Negative Pressure Wound Therapy | Standard Dressing
Number analyzed (Participants) | 37 | 42
Participants
  chorioamnionitis | 4 | 3
  no chorioamnionitis | 33 | 39
Statistical Analysis 1: Comparison: Negative Pressure Wound Therapy vs Standard Dressing; Test type: Other — Cochran-Mantel-Haenzel measure used to estimate interaction between chorioamnionitis and no chorioamnionitis stratified by icNPT and standard dressing, for wound morbidity; p = 0.74, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: 1 year, 8 months
Arm/Group | Negative Pressure Wound Therapy | Standard Dressing
All-Cause Mortality (participants affected / at risk) | 0/222 | 0/219
Serious Adverse Events (participants affected / at risk) | 0/222 | 0/219
Other Adverse Events (participants affected / at risk) | 0/222 | 0/219

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
8. PUBLICATION AND REPORTS ON DATA; COPYRIGHTS

A. Prior to public presentation or submission to a journal, Investigator will submit for review to Company...content of any manuscript for publication, abstract, or presentation containing data and results of the Study, ...such review is for the limited purposes of ensuring that the manuscript accurately describes the Product and does not contain any Confidential lnformation...Investigator will have the unfettered right to publish.